CLINICAL TRIAL: NCT06834711
Title: Chlorhexidin Versus N-Asetil Sistein Irrigation in Mandibular Molar Teeth with Chronic Apical Periodontitis on Postoperative Pain and Periapical Tissue Healing: a Randomized Controlled Trial
Brief Title: Chlorhexidine Versus N-Asetil Sistein Irrigation in Mandibular Molar Teeth with Chronic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Cukurova University, Faculty of Dentistry, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13.02.2025/152
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chronic Apical Periodontitis
Keywords: chronic apical periodontitis; postoperative pain; N-asetil sistemin; chlorhexidin
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetylcysteine; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): During root canal preparation, each canal was irrigated with a total of 18 ml of 2.5% sodium hypochlorite (NaOCl). In the final irrigation, each root canal was irrigated with 3 ml of 17% ethylene diamine tetra-acetic acid (EDTA) for 1 minute, followed by 5 ml of distilled water. Then, 5 ml of 2.5% NaOCl was irrigated, and finally 5 ml of distilled water was used.
- Chlorhexidine Group (Experimental): During root canal preparation, each canal was irrigated with a total of 18 ml of 2.5% NaOCl. In the final irrigation, each root canal was irrigated with 3 ml of 17% ethylene diamine tetra-acetic acid (EDTA) for 1 minute, followed by 5 ml of distilled water. Then, each canal was irrigated with 3 ml of 2% chlorhexidine (CHX) and finally 5 ml of distilled water was used.
  Interventions: Drug: Chlorhexidine
- N-asetil Sistein Group (Experimental): During root canal preparation, each canal was irrigated with a total of 18 ml of 2.5% NaOCl. In the final irrigation, each root canal was irrigated with 3 ml of 17% ethylene diamine tetra-acetic acid (EDTA) for 1 minute, followed by 5 ml of distilled water. Then, each canal was irrigated with 3 ml of N-acetyl Cysteine (NAC) (200 mg/ml) and finally 5 ml of distilled water was used.
  Interventions: Drug: N-Acetyl Cysteine

INTERVENTIONS:
Drug: N-Acetyl Cysteine — The root canals were irrigated with 3 mL N-acetyl Cysteine (NAC)(200 mg/ml) in N-acetyl Cysteine group in the final irrigation.
  Arms: N-asetil Sistein Group
Drug: Chlorhexidine — The root canals were irrigated with 3 ml %2 chlorhexidine in chlorhexidin group in the final irrigation.
  Arms: Chlorhexidine Group

SUMMARY:
The goal of this clinical study was to evaluate the effect of using different irrigation solutions in the final irrigation of root canal treatment procedures on the intensity of postoperative pain and periapical tissue healing in patients presenting with mandibular molars with chronic apical periodontitis. The main question it aims to answer is:

- Does controlled irrigation with chlorhexidin and N-asetil sistein in root canal treatment reduce the severity of postoperative pain? In the chlorhexidin group, unlike the control group, each root canal was irrigated with 3 mL %2 chlorhexidin solution in the final irrigation.

In the N-asetil sistein group, unlike the control group, each root canal was irrigated with 3 mL 200 mg/ml N-asetil sistein solution in the final irrigation.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular permanent molars with chronic apical periodontitis
* Teeth with periapical index (PAI) score greater than 2
* Teeth with periodontal pocket depth less than 3 mm
* Patients without systemic disease (ASA 1-2)

Exclusion Criteria:

* Patients who have used analgesic, anti-inflammatory or opioid drugs in the last 7 days or antibiotics in the last 3 months
* Patients who report pregnancy, lactation or psychiatric disorders
* Teeth with a history of root canal treatment, sinus tract or abscess, and teeth planned for prosthetic restoration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corazza BJM, Martinho FC, Khoury RD, Toia CC, Orozco EIF, Prado RF, Machado FP, Valera MC. Clinical influence of calcium hydroxide and N-acetylcysteine on the levels of resolvins E1 and D2 in apical periodontitis. Int Endod J. 2021 Jan;54(1):61-73. doi: 10.1111/iej.13403. Epub 2020 Oct 3. PMID 32896000
- [Background] Comparative evaluation of N-acetylcysteine and chlorhexidine as final irrigation on the push-out bond strength of different sealers: An in vitro study